CLINICAL TRIAL: NCT01459445
Title: Metformin Plus EE30µg-drospirenone and Weight Loss- Impact on Endothelial Function and hsCRP Levels in PCOS
Brief Title: Metformin+ Drospirenone/ethinylestradiol30µg and Flow-mediated Dilation in Polycystic Ovary Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Iuliu Hatieganu University of Medicine and Pharmacy (Other)
Responsible Party: Principal Investigator, Carmen Georgescu, Associated Professor, Iuliu Hatieganu University of Medicine and Pharmacy
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IuliuHatieganuU246; PNCDI II 41_068/2007 (Other Grant/Funding Number: Romanian Ministry of Education and Research)
Record Dates: First submitted 2011-10-18; First posted 2011-10-25 (Estimated); Last update posted 2011-10-25 (Estimated); Status verified 2011-10

CONDITIONS: Polycystic Ovary Syndrome; Endothelial Dysfunction
Keywords: ethinylestradiol 30µg-drospirenone; flow-mediated dilatation; endothelial dysfunction; hsCRP; metformin; polycystic ovary syndrome
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Metformin; Ethinyl Estradiol; drospirenone; drospirenone and ethinyl estradiol combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Metformin+Drospirenone / EE 30µg (Other)
  Interventions: Drug: Metformin, Ethinylestradiol 30µg-Drospirenone

INTERVENTIONS:
Drug: Metformin, Ethinylestradiol 30µg-Drospirenone — Metformin: 1700 mg /day (twice per day)-6 months; EE30µg-drospirenone: 1 tb/day, 21 days/month, 6 months
  Other Names: metformin; yasmin

SUMMARY:
The purpose of this study is to assess the effects of ethinylestradiol 30µg-drospirenone combined with metformin and weight loss by means of dietary intervention on the indices of endothelial dysfunction (i.e. flow-mediated dilation and serum endothelin-1), serum hsCRP,lipids,insulin resistance and body composition in young women with PCOS.

DETAILED DESCRIPTION:
Women with polycystic ovary syndrome (PCOS) frequently cluster several cardiovascular risk markers and early subclinical atherosclerosis. Because combined oral contraceptives (COCs), the most common treatment of this disease, might adversely influence insulin resistance, glucose tolerance, lipid profile or aggravate chronic inflammation the possibility of worsening the already unfavorable cardiovascular risk profile of PCOS subjects is of concern. On the contrary, the insulin sensitizer metformin has been shown to ameliorate insulin resistance, reduce hyperandrogenism and triglyceride levels and also to improve endothelial structure and function in PCOS. Drospirenone (DRP) is a progestin with antiandrogenic and antimineralocorticoid activity. However, the studies assessing the effect of the COC containing 30 µg EE+3mg DRP (DRP/EE30µg) on surrogate markers of atherosclerosis are few and inconclusive. Therefore,the purpose of the present study is to assess the effects of the oral contraceptive DRP/EE30µg combined with metformin and weight loss by means of dietary intervention on the indices of endothelial dysfunction, i.e. flow-mediated dilation and serum endothelin-1, serum hsCRP,lipids, and insulin resistance in young women with PCOS.

ELIGIBILITY:
Inclusion Criteria:

* women with diagnosis of polycystic ovary syndrome defined according to Androgen Excess Society 2006 guidelines

Exclusion Criteria:

* secondary causes of hyperandrogenism such as hyperprolactinemia, thyroid disease, androgen-secreting tumours, Cushing's syndrome and congenital adrenal hyperplasia
* current or previous use (within 6 months) of oral contraceptives, anti-androgens, ovulation induction medications
* use of drugs known to affect carbohydrate-lipid metabolism or inflammation (anti-inflammatory drugs) at the time of evaluation and during the last one month preceding the evaluations
* concurrent minor infection reported during the last one month preceding the evaluations
* personal history of diabetes mellitus

Ages: 15 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 26 (Estimated)
Dates: Start 2011-02; Primary Completion 2011-06 (Actual); Study Completion 2012-01 (Estimated)

PRIMARY OUTCOMES:
flow-mediated dilation | six months

SECONDARY OUTCOMES:
endothelin-1 | six months
hsCRP | six months
insulin resistance indices | six months
body composition | six months
lipid profile | six months
total testosterone | six months
sex hormone-binding globulin | six months
systolic blood pressure and diastolic blood pressure | six months

CONTACTS AND LOCATIONS:
Overall Officials: Carmen Georgescu, Principal Investigator — University of Medicine and Pharmacy Iuliu Hatieganu
Locations (1):
- Clinic of Endocrinology, Cluj-Napoca, Cluj, Romania

REFERENCES:
- [Derived] Ilie IR, Marian I, Mocan T, Ilie R, Mocan L, Duncea I, Pepene CE. Ethinylestradiol30mug-drospirenone and metformin: could this combination improve endothelial dysfunction in polycystic ovary syndrome? BMC Endocr Disord. 2012 Jun 19;12:9. doi: 10.1186/1472-6823-12-9. PMID 22713099